CLINICAL TRIAL: NCT00087191
Title: Distribution Of The Photosensitizer Motexafin Lutetium And Hypoxia In Patients With Malignancies
Brief Title: EF5 and Motexafin Lutetium in Detecting Tumor Cells in Patients With Abdominal or Non-Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI-2012-02607; UPCC# 04204; P01CA087971 (NIH); CDR0000373812 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Adult Primary Liver Cancer; Carcinoma of the Appendix; Fallopian Tube Cancer; Gastrointestinal Stromal Tumor; Localized Extrahepatic Bile Duct Cancer; Localized Gallbladder Cancer; Localized Gastrointestinal Carcinoid Tumor; Localized Resectable Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Metastatic Gastrointestinal Carcinoid Tumor; Ovarian Sarcoma; Ovarian Stromal Cancer; Primary Peritoneal Cavity Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Adult Soft Tissue Sarcoma; Recurrent Colon Cancer; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Recurrent Gastric Cancer; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Recurrent Small Intestine Cancer; Recurrent Uterine Sarcoma; Regional Gastrointestinal Carcinoid Tumor; Small Intestine Adenocarcinoma; Small Intestine Leiomyosarcoma; Small Intestine Lymphoma; Stage 0 Non-small Cell Lung Cancer; Stage I Adult Soft Tissue Sarcoma; Stage I Colon Cancer; Stage I Gastric Cancer; Stage I Non-small Cell Lung Cancer; Stage I Ovarian Epithelial Cancer; Stage I Ovarian Germ Cell Tumor; Stage I Pancreatic Cancer; Stage I Rectal Cancer; Stage I Uterine Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage II Colon Cancer; Stage II Gastric Cancer; Stage II Non-small Cell Lung Cancer; Stage II Ovarian Epithelial Cancer; Stage II Ovarian Germ Cell Tumor; Stage II Pancreatic Cancer; Stage II Rectal Cancer; Stage II Uterine Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage III Colon Cancer; Stage III Gastric Cancer; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage III Pancreatic Cancer; Stage III Rectal Cancer; Stage III Uterine Sarcoma; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Adult Soft Tissue Sarcoma; Stage IV Colon Cancer; Stage IV Gastric Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Stage IV Uterine Sarcoma; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Appendiceal Neoplasms; Fallopian Tube Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Sarcoma; Colonic Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Rectal Neoplasms | interventions — motexafin lutetium

ARMS (1):
- Diagnostic (EF5, motexafin lutetium) (Experimental): Patients receive EF5 IV over 1-2.5 hours on day 1 and motexafin lutetium IV over 10-15 minutes on day 2. Patients undergo definitive surgical resection approximately 3 hours after motexafin lutetium administration. Hypoxia and motexafin lutetium levels in the resected tumors are evaluated. Tumor to normal tissue ratios are also determined.
  Interventions: Drug: EF5; Drug: motexafin lutetium; Other: pharmacological study

INTERVENTIONS:
Drug: EF5 — Given IV
Drug: motexafin lutetium — Given IV
  Other Names: Antrin; lutetium texaphrin; lutetium texaphyrin; Lutex; PCI-0123
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This clinical trial is studying the amount of EF5 and motexafin lutetium present in tumor cells and/or normal tissues of patients with abdominal (such as ovarian, colon, or stomach cancer) or non-small cell lung cancer. EF5 may be effective in measuring oxygen in tumor tissue. Photosensitizing drugs such as motexafin lutetium are absorbed by tumor cells and, when exposed to light, become active and kill the tumor cells. Knowing the level of oxygen in tumor tissue and the level of motexafin lutetium absorbed by tumors and normal tissue may help predict the effectiveness of anticancer therapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the uptake of motexafin lutetium in tumors and normal tissue of patients with intra-abdominal malignancies or non-small cell lung cancer.

II. Determine the ratio of tumor to normal tissue by measuring the level of motexafin lutetium uptake in tumor and normal tissue removed from these patients.

III. Determine the pattern, presence, and level of EF5 binding (as a surrogate marker for hypoxia) in tumors of these patients.

IV. Determine the feasibility of measuring optical properties, tissue oxygenation, motexafin lutetium concentration, fluorescence, and blood flow by non-invasive means in these patients.

OUTLINE: This is a multicenter, diagnostic study. Patients are stratified according to diagnosis (intra-abdominal malignancy vs non-small cell lung cancer).

Patients receive EF5 IV over 1-2.5 hours on day 1 and motexafin lutetium IV over 10-15 minutes on day 2. Patients undergo definitive surgical resection approximately 3 hours after motexafin lutetium administration. Hypoxia and motexafin lutetium levels in the resected tumors are evaluated. Tumor to normal tissue ratios are also determined.

After completion of study treatment, patients are followed at approximately 1-8 weeks.

PROJECTED ACCRUAL: A total of 30 patients (20 with intra-abdominal malignancies and 10 with non-small cell lung cancer) will be accrued for this study within 10-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or suspected diagnosis of 1 of the following:

  * Intra-abdominal malignancy of 1 of the following types:

    * Sarcoma
    * Ovarian cancer
    * Gastrointestinal malignancies, including, but not limited to, appendiceal cancer, colon cancer, or gastric cancer
  * Non-small cell lung cancer
* Planning to undergo surgical resection of disease
* Disease has the propensity to spread to the peritoneal cavity (intra-abdominal malignancy patients)
* Performance status - ECOG 0-2
* WBC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin < 1.5 mg/dL
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* Body weight ≤ 130 kg
* No G6PD deficiency
* No porphyria
* No history of peripheral neuropathy ≥ grade 3
* Able to tolerate anesthesia and major surgery
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Motexafin lutetium uptake in tumors and normal tissues | At the time of surgery
  Data will be described using graphical techniques (e.g., box plots) and summary statistics (e.g., means, medians, standard deviations, and interquartile ranges). For each patient, the mean concentration of motexafin lutetium across tumor and normal samples will be summarized.
Tumor to normal tissue ration (TNTR) of motexafin lutetium for any tumor and normal tissue | At the time of surgery
  Summary data for each patient will be used to construct a TNTR. Wilcoxon signed rank test of whether the median ration exceeds will be carried out.
Pattern and presence of EF5 binding | At the time of surgery
  EF5 biding will be quantified.
Toxicity as assessed by NCI Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 60 days following EF5 infusion
  Will be graded, tabled for each stratum and for the entire study and summarized by frequencies and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States